CLINICAL TRIAL: NCT05603754
Title: A Phase 3, 16-Week, Multicenter, Randomized, Double Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of a Single Injection of Lorecivivint 0.07 mg Dose in the Target Knee Joint of Subjects With Moderate to Severe Osteoarthritis Pain of the Knee
Brief Title: A Study Utilizing Patient-Reported Outcomes to Evaluate the Safety and Efficacy of Lorecivivint (SM04690) for the Treatment of Moderately to Severely Symptomatic Knee Osteoarthritis (STRIDES)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biosplice Therapeutics, Inc. (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SM04690-OA-21
Record Dates: First submitted 2022-10-27; First posted 2022-11-03 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — lorecivivint

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lorecivivint (Experimental): Healthcare professional-administered intra-articular injection; performed on Day 1.
  Interventions: Drug: Lorecivivint
- Vehicle (Placebo Comparator): Healthcare professional-administered intra-articular injection; performed on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lorecivivint — One intra-articular injection of 0.07 mg lorecivivint in 2 mL vehicle
  Other Names: SM04690
  Arms: Lorecivivint
Drug: Placebo — One intra-articular injection of 0 mg lorecivivint in 2 mL vehicle
  Other Names: Vehicle
  Arms: Vehicle

SUMMARY:
This phase 3 study is a multicenter, randomized, double-blind, placebo-controlled study of lorecivivint injected intra-articularly (IA) into the target (most painful) knee joint of moderately to severely symptomatic osteoarthritis (OA) subjects at a single dose of 0.07 mg lorecivivint per 2 mL injection. This study will utilize standard outcomes to evaluate the safety and efficacy of lorecivivint.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 40 and 80 years of age, inclusive, in general good health apart from their knee OA
* Ambulatory (single assistive devices such as canes allowed if needed less than 50% of the time, subjects requiring a walker are excluded)
* Diagnosis of femorotibial OA in the target knee by standard American College of Rheumatology (ACR) criteria at the Screening Visit (clinical AND radiographic criteria); OA of the knee is not to be secondary to any rheumatologic conditions (e.g., rheumatoid arthritis)
* Radiographic disease Stage 2 or 3 in target knee within 24 weeks of the Screening Visit according to the Kellgren-Lawrence (KL) grading of knee OA as assessed by independent central readers
* Qualifying mean score on the 24-h average pain score (0-10 numeric rating scale)
* Pain compatible with OA of the knee(s) for at least 26 weeks prior to the Screening Visit
* Primary source of pain throughout the body is due to OA in the target knee
* Body mass index (BMI) ≤ 35 kg/m2 at the Screening Visit

Exclusion Criteria:

* Pregnant women, breastfeeding women, and women who are not post-menopausal (defined as 12 months with no menses without an alternative medical cause) or permanently surgically sterile (includes hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) who have a positive or indeterminate pregnancy test result at the Screening Visit or Day 1
* Partial or complete joint replacement in either knee
* Currently requires use of a lower extremity prosthesis, and/or a structural knee brace (i.e., a knee brace that contains hardware)
* Any surgery (e.g., arthroscopy) in either knee within 26 weeks prior to Day 1
* Intra-articular (IA) injection into the target knee with a therapeutic aim including, but not limited to hyaluronic acid, platelet-rich plasma (PRP), and stem cell therapies within 26 weeks prior to Day 1; or IA glucocorticoids within 12 weeks prior to Day 1 allowed
* Previous treatment with lorecivivint (SM04690)
* Participation in a clinical research trial that included the receipt of an investigational product or any experimental therapeutic procedure within 26 weeks prior to the Screening Visit, or planned participation in any such trial
* Subjects requiring the use of opioids > 1x per week within 12 weeks prior to Day 1
* History of malignancy within the last 5 years; not including subjects with prior history of adequately treated in situ cervical cancer or basal or squamous cell skin cancer
* Clinically significant abnormal screening hematology values, blood chemistry values, or urinalysis values as determined by the Investigator
* Any known active infections, including urinary tract infection, upper respiratory tract infection, sinusitis, suspicion of IA infection, hepatitis B or hepatitis C infection, and/or infections that may compromise the immune system such as human immunodeficiency virus (HIV) at Day 1
* Use of APAP or NSAIDs during washout period (between Screening Visit 2 and Day 1). Use of aspirin (up to 325 mg/day) for thrombosis prophylaxis is permitted.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline OA pain in the target knee as assessed by weekly average of daily pain numeric rating scale (NRS) at Week 12 | Baseline and Week 12
  Evaluate change from baseline OA pain in the target knee as assessed by weekly average of daily pain NRS at Week 12. The pain NRS is an 11-point scale [0-10] for subject self-reporting of average knee pain in the last 24 hours; 0 indicates no pain, and 10 indicates pain as bad as you can imagine.

SECONDARY OUTCOMES:
Change from baseline OA function as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) physical function subscore (WOMAC Function) at Week 12 | Baseline and Week 12
  Evaluate change from baseline OA function as assessed by WOMAC Function at Week 12. The WOMAC is a widely-used, proprietary outcome measurement tool used to evaluate the condition of subjects with OA of the knee and hip, including pain (5 questions), stiffness (2 questions) and physical functioning (17 questions) of the joints. Each question is measured on an 11-point NRS scale [0-10]; 0 indicates no pain / no stiffness / no difficulty, and 10 indicates extreme pain / extreme stiffness / extreme difficulty. The WOMAC Function subscore is scaled to range from 0 to 100.
Change from baseline OA disease activity as assessed by Patient Global Assessment at Week 12 | Baseline and Week 12
  Evaluate change from baseline OA disease activity as assessed by Patient Global Assessment at Week 12. The Patient Global Assessment is an 11-point NRS [0-10] for subject self-reporting of how they feel their target knee is impacting them; 0 indicates very good, and 10 indicates very bad.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Yazici, MD, Study Director — Biosplice Therapeutics, Inc.
Locations (43):
- United States (43):
  - Tucson Orthopaedic Institute, Tucson, Arizona
  - Core Healthcare Research, Cerritos, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Infinity Clinical Research, Norco, California
  - Dream Team Clinical Research, Pomona, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Millennium Clinical Trials, LLC, Thousand Oaks, California
  - Unique Clinical Trials, Doral, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - TecTum Research, Hollywood, Florida
  - Columbus Clinical Services, LLC, Miami, Florida
  - AppleMed Research Group, LLC, Miami, Florida
  - Advance Medical Research Center, Miami, Florida
  - Health and Life Research Institute, LLC, Miami, Florida
  - BioMed Research and Medical Center, Miami, Florida
  - Well Pharma Medical Research, Corp, Miami, Florida
  - South Florida Research Phase I-IV, Inc., Miami Springs, Florida
  - Tampa Pain Relief Center, Tampa, Florida
  - Premier Medical Associates, The Villages, Florida
  - Conquest Research, LLC, Winter Park, Florida
  - Pinnacle Trials, Inc., Stockbridge, Georgia
  - Chicago Clinical Research Institute, Chicago, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - DelRicht Research - Mandeville, Mandeville, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - DelRicht Research - Prairieville, Prairieville, Louisiana
  - DelRicht Research - Rockville, Rockville, Maryland
  - Skylight Health Research, Burlington, Massachusetts
  - Oakland Medical Research, Troy, Michigan
  - Healthcare Research Network, Hazelwood, Missouri
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Hightop Medical Research Center, Cincinnati, Ohio
  - Conrad Clinical Research, Edmond, Oklahoma
  - DelRicht Research - Tulsa, Tulsa, Oklahoma
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Piedmont Research Partners, LLC, Fort Mill, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Zenos Clinical Research, Dallas, Texas
  - Synergy Groups Medical, LLC, Houston, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Diagnostic Research Group, San Antonio, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah